CLINICAL TRIAL: NCT04543253
Title: Recovery From Cushing Syndrome and Mild Autonomous Cortisol Secretion (MACS)
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Irina Bancos, Principal Investigator, Mayo Clinic
Other Study IDs: 19-006003
Record Dates: First submitted 2020-04-10; First posted 2020-09-10 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Cushing Syndrome
Keywords: Hypercortisolism; Cushing syndrome; Cushing disease; Pituitary
MeSH Terms: conditions — Cushing Syndrome; Pituitary ACTH Hypersecretion; Pituitary Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Standard of care CS: Patients undergoing curative surgery for any type of CS who will be followed through standard of care after surgery
- MUSE intervention CS: Patients undergoing curative surgery for any type of CS who will be introduced to and provided MUSE for use after surgery
  Interventions: Other: MUSE biofeedback

INTERVENTIONS:
Other: MUSE biofeedback — biofeedback through a headband
  Groups: MUSE intervention CS

SUMMARY:
Cushing syndrome (CS) is an endocrine disorder caused by chronic exposure to glucocorticoid (GC) excess. Endogenous CS has an estimated incidence of 0.2 to 5.0 cases per million per year and prevalence of 39 to 79 cases per million in various populations. CS usually affects young women, with a median age at diagnosis of 41.4 with a female-to-male ratio of 3:1. Following a curative surgery for CS, patients develop adrenal insufficiency and require GC replacement postoperatively until the hypothalamic-pituitary-adrenal (HPA) axis recovery occurs. Factors, such as age, gender, BMI, subtypes of CS, duration of symptoms, clinical and biochemical severity and postoperative GC dose have been reported to affect the HPA recovery in small retrospective studies. Glucocorticoid withdrawal syndrome (GWS) is a withdrawal reaction due to decrease in supraphysiological GC concentrations, which occurs after a successful surgery of CS. Glucocorticoid withdrawal syndrome (GWS) is under-recognized entity in patients undergoing curative surgery for endogenous Cushing syndrome.

In this study we aim to determine pre- and post-surgical predictors of the duration and severity of glucocorticoid withdrawal in patients undergoing a curative surgery for cortisol excess and assess the effect of MUSE intervention on GWS severity in patients undergoing curative surgery for CS as compared to standard of care.

DETAILED DESCRIPTION:
Specific Aim 1: To determine pre- and post-surgical predictors of the duration and severity of glucocorticoid withdrawal in patients undergoing a curative surgery for cortisol excess Specific Aim 2: To characterize the timing and recovery of hypercortisolism-induced signs and symptoms, proximal myopathy and tissue accumulation of Advanced Glycation End products (AGEs) in patients after a curative surgery Specific Aim 3: To assess the effect of MUSE intervention on GWS severity in patients undergoing curative surgery for CS as compared to standard of care

1. Selection of study subjects and medical records review. We will prospectively recruit adult patients with CS of any three subtypes (pituitary, adrenal or ectopic CS) and MACS undergoing a curative surgery, from the pituitary clinic. Investigator will discuss participation in the study and obtain an informed consent. We will review data for any potential risk factors through clinical interview and review of medical record. Data will include demographics, behavioral factors (smoking and alcohol consumption), past medical history (history of AI, psychiatric disorder and recent GC usage), GWS related symptoms and signs (anorexia, nausea, emesis, lethargy, somnolence, arthralgia, myalgia, fever, hypotension), and lab tests.
2. Subjects: We will enroll 100 consecutive subjects in this study who will participate in this study for up to 2 years. Inclusion and exclusion criteria are as below. We plan to have 50 subjects participate in the intervention arm with MUSE in one year, without modifying other study procedures.
3. Step-by-Step methods:

   * Patients will be identified by their clinician. Permission will be obtained from the patient in order for one of the investigators to explain the study and obtain informed written consent.
   * Baseline history, physical examination, and the necessary baseline tests will be performed based on standard of care and as considered necessary by the treating physician.
   * Medical record will be reviewed for demographic information, comorbidities, medical therapy, imaging information and biochemical testing results
   * We will use a scoring system to quantify biochemical severity, and to classify clinical abnormalities as mild, moderate and severe ( based on existent laboratory and clinical parameters).
   * At baseline, all patients will be asked to complete the Cushing QoL questionnaire, SF36 and AddiQol questionnaires (forms are attached in Document). Patients will discuss the intervention with MUSE with the study investigator. If they agree to participate in the intervention arm, they will be instructed on its use.
   * At follow up, patients will complete AddQoL survey (weekly in the first 3 months, every 4 weeks in the next 6 months, every 3 months in the next 12 months, and then every 6 months until the end of the study) and SF36 survey (every 3 months) until the end of the study. (In-person, through a paper survey or electronically using external REDCap server (user name and password protected)).
   * For patients in the intervention group, in addition to the above, at the time of enrollment, the study coordinator will help set up the MUSE application on to iPad or iPhone or Android phone (we will use generic login name and password without protected health information included). The coordinator will also go over a few helpful hints and discuss the homework log, which will need to be completed throughout the course of the study. After the surgery, patients are asked to complete the 3 minute 'focusing' exercise daily until 12 weeks after the surgery. During this time frame we will download the data from our end on a weekly basis. After 12 weeks, the frequency of the usage will be at the participant's discretion although ongoing usage is encouraged and data download should continue. In addition, we ask that patients bring iPad, iPhone or Android phone to each of the clinical visit for an app interrogation.
   * Patient will participate in the study until one of the following: 1) 2 years of follow up completed, 2) patient withdraws consent, 3) HPA axis recovery is achieved and patient weans off GC, 4) completion of the study by the principal investigator.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 and above,
2. new diagnosis of CS of any of the three subtypes (pituitary, adrenal or ectopic CS), and MACS,
3. planning for a curative surgery
4. ability to provide informed consent.

Exclusion Criteria:

1. systemic supraphysiological GC for any reason within 1 month of enrollment, for more than 2 weeks,
2. inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any male or female at least 18 years of age undergoing curative surgery for Cushing's Syndrome and MACS.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2019-07-25 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Quality of life (SF36) | periodic 0-24 months
  Score 0-100

SECONDARY OUTCOMES:
HPA recovery | 0-24 months
  as measured by morning cortisol. Cortisol measurement will be performes every 6-12 weeks, 24h off glucocorticoid replacement therapy starting 4 weeks-8 weeks after surgery and until cortisol is 10 mcg/dl or above ( or HPA recovery is considered impossible by investigator)
Myopathy measurement | 0-24 months
  as measured by hand grip. Hand grip strength will be measured 3 times on left and right, and dominant hand grip strength will be considered as an average of 3 measurements.

OTHER OUTCOMES:
AGE | 0-24 months
  measurement of AGE

CONTACTS AND LOCATIONS:
Overall Officials: Irina Bancos, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials